CLINICAL TRIAL: NCT07385690
Title: Xpan Non-Inferiority Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Lawrence Tabone, Associate Professor and Chief of Division of General Surgery, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2506178705
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Xpan Trocar System (Active Comparator): Participants will undergo laparoscopic surgery using the Xpan Trocar System. Standard insertion technique will be used to create a 3 mm punch into an already gas-extended abdomen. A total of 3-5 trocars will be placed based on the type of surgery. Once placed, trocars will be radially dilated to the size necessary for the procedure, generally 2 trocars expanded to 5 mm and 2 trocars expanded to 12 mm. Final trocar size will range from 3 mm to 12 mm. Both placement and final dilated size will be documented.
  Interventions: Device: Xpan Trocar System
- Standard of Care (Non-expanding Trocar) (Placebo Comparator): Participants will undergo laparoscopic surgery using a non-expanding trocar, which is considered the institutions standard of care for the procedure. Trocar size is selected based on surgical requirements and remain fixed throughout the procedure.
  Interventions: Device: Standard of Care (Non-expanding Trocar)

INTERVENTIONS:
Device: Xpan Trocar System — A radially dilating trocar system intended to reduce incision trauma by gradually dilating tissue rather than cutting. Allows initial placement at 3 mm and expansion up to 12 mm as needed for surgical access.
  Arms: Xpan Trocar System
Device: Standard of Care (Non-expanding Trocar) — A surgical access device used during laparoscopic procedures that does not expand the incision site and is routinely used in standard practice.
  Arms: Standard of Care (Non-expanding Trocar)

SUMMARY:
A trocar is a surgical instrument with a sharp point and tube and is used to create endoscopic access in the abdomen or chest where endoscopic instruments can be entered & used in minimally invasive surgical procedures. Xpan has created an FDA Cleared radially dilating trocar (RDT) that is inserted at 3mm and can be expanded to 5mm or 12mm during surgery. The purpose of this research protocol is to demonstrate that a new FDA Cleared Xpan® radially dilating trocar (RDT) system is at least, just as effective as the existing RDT trocar systems. The procedure will be performed using a radially dilating trocar that is inserted at 3mm and can be expanded to 5mm or 12mm during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals scheduled for the following procedures:

  * Sleeve Gastrectomy
  * Bypass
  * Revision & other bariatric procedures
  * Robotic procedures
  * Bariatric patients

Exclusion Criteria:

* Any individual not scheduled for the above procedure and/or does not meet the age requirments.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Trocar slippage and Displacement | Day 1- At time of procedure
  Percentage of trocars inserted for use during surgery that need to be adjusted or reinserted during surgical procedure due to slippage and/or displacement.

SECONDARY OUTCOMES:
Percentage of Cases Without Fascial Closure at 12 mm Sites | Day 1- At time of procedure
  The proportion of surgical cases where fascial closure was not required at 12 mm trocar sites.
Incidence of Trocar-Related Complications | Day 1- At time of procedure
  The number of trocar-related complications (e.g., bleeding, infection, loss of pneumoperitoneum) observed during surgery.
Ease of Use of Expansion Technique | Day 1- At time of procedure
  Surgeon-reported ease of use of the trocar expansion technique, rated on a 1-5 Likert scale (1 = difficult to use, 5 = easy to use) with 5 being the best outcome.
Frequency of Trocar Upsizing | Day 1- during procedure
  The percentage of trocar insertions requiring upsizing.
Surgeon reported Ease of Trocar Upsizing | Day 1- during procedure
  The surgeon-reported ease of upsizing, rated on a 1-5 Likert scale (1 = difficult, 5 = easy) with 5 being the best outcome.
Percentage that Maintained Abdominal Pathway and Pneumoperitoneum During Upsizing | Day 1- At time of procedure
  Percentage of successful maintenance of abdominal pathway and pneumoperitoneum during trocar upsizing.
Total Procedure Time | Day 1- At time of procedure
  Total time (in minutes) from insufflation and trocar insertion to completion of the surgical procedure.
Postoperative Analgesic Use | Up to 72 hours post procedure
  Percentage of participants reporting postoperative analgesic consumption.
Time to Return to Normal Activity | 6 weeks post procedure
  Number of days until return to work or normal activity.
Postoperative Pain Scores | 4 hours post procedure
  Pain scores measured postoperatively using a standardized pain scale (e.g., 0-10 Numeric Rating Scale) with 10 being the worst pain/outcome.
Postoperative Pain Scores | 8 hours post procedure
  Pain scores measured postoperatively using a standardized pain scale (e.g., 0-10 Numeric Rating Scale) with 10 being the worst pain/outcome.
Postoperative Pain Scores | 12 hours post procedure
  Pain scores measured postoperatively using a standardized pain scale (e.g., 0-10 Numeric Rating Scale) with 10 being the worst pain/outcome.
Postoperative Pain Scores | 24 hours post procedure
  Pain scores measured postoperatively using a standardized pain scale (e.g., 0-10 Numeric Rating Scale) with 10 being the worst pain/outcome.
Postoperative Pain Scores | 72 hours post procedure
  Pain scores measured postoperatively using a standardized pain scale (e.g., 0-10 Numeric Rating Scale) with 10 being the worst pain/outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Tabone, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No